CLINICAL TRIAL: NCT00113152
Title: Are Left Ventricular Abnormalities Associated With Pulmonary Hypertension in Sickle Cell Anemia?
Brief Title: Heart Disease in Sickle Cell Anemia
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 050154; 05-CC-0154
Record Dates: First submitted 2005-06-03; First posted 2005-06-06 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2007-10-02

CONDITIONS: Sickle Cell Anemia; Pulmonary Hypertension
Keywords: Cardiac Arrhythmias; Diastolic Dysfunction; Pulmonary Hypertension; Sickle Cell Anemia; Sudden Death; Thalassemia
MeSH Terms: conditions — Anemia, Sickle Cell; Hypertension, Pulmonary; Arrhythmias, Cardiac; Death, Sudden; Thalassemia

SUMMARY:
This study will explore what may cause people with sickle cell anemia to have heart problems and an increased risk of sudden death.

People 18 years of age and older with sickle cell anemia may be eligible for this study. Candidates are screened with a medical history and physical examination, electrocardiogram (EKG), echocardiogram (heart ultrasound), and blood tests.

Participants undergo the following tests and procedures:

* Holter monitoring: The patient wears a small, battery-operated device to record heart rate and rhythm over 24 to 48 hours.
* QRST surface mapping: An EKG using 64 electrodes is done at rest and during exercise to provide a detailed look at the heart and its conduction system.
* Chest x-rays are taken to examine the lungs.
* Bicycle exercise echocardiography test: Blood pressure, pulse, heart rhythm and oxygen use are monitored while the patient exercises on a stationary bicycle. Ultrasound pictures are also obtained during the exercise.
* Echocardiogram: A heart ultrasound is done to check how well the heart is pumping blood.
* Pulmonary artery catheterization: A catheter (plastic tube) is inserted into a vein and advanced to the chambers of the heart, through the heart valve and into the lung artery. The pressures in the heart and lung blood vessels are measured while the patient is resting and during exercise, with the bed tilted up and down, and after giving 500 mls of fluid into a vein.
* Blood tests are done to measure a hormone called brain natriuretic peptide, which can increase with the development of heart failure, and nitrite, a substance that can affect blood vessel dilation. Some blood is stored to test for inflammatory markers and for possible future gene and protein analysis.
* Cardiac magnetic resonance imaging (cMRI): The patient lies in a donut-shaped magnet while pictures of the heart are obtained using a magnetic field and radio waves. Earplugs are worn to muffle the loud sounds that occur with electrical switching of the magnetic fields. A contrast agent called gadolinium may be injected to enhance the quality of the images.
* Invasive electrocardiographic (reveal) monitoring: This procedure permits study of the heart rhythms over a long time period. A small device is placed just under the skin on the left side of the chest. It can be left in for up to 14 months to monitor the heartbeat continuously during this time.

DETAILED DESCRIPTION:
Sickle cell anemia is an inherited blood disorder primarily affecting groups with origins in endemic malarial areas, especially those of African descent. SCA results from one of two single amino-acid substitutions in beta-hemoglobin (Hb-S and Hb-C) that increases the propensity for hemoglobin to polymerize, thus distorting, sickling and hemolyzing red cells. Individuals homozygous for Hb-S (or double heterozygote Hb-S and Hb-C) develop sickle cell anemia (SCA), while heterozygotes have sickle cell trait. SCA is characterized by chronic anemia and crises of red cell sickling and ischemia that are often painful and affect several organs and tissue types. SCA confers considerable disability, morbidity and mortality.

Annual mortality from SCA has been estimated at approximately 3%. As a significant number of these deaths are sudden, a cardiac cause has been suspected. However, no cardiac mechanism of sudden death (SD) has been clearly identified. Recently, it has been demonstrated that SCA patients with pulmonary hypertension (PAH) have a higher incidence of SD than those with normal pulmonary pressures. In many patients, PAH occurs in association with elevated pulmonary arterial wedge pressures and normal pulmonary arterial resistance, suggesting that the PAH develops as the result of left ventricular (LV) abnormalities. Furthermore, in other conditions in which PAH develops, SD occurs only at pressures considerably higher than those observed in SCA. These factors suggest that PAH in SCA is a surrogate marker for, rather than the cause of SD. Rather, an SCA cardiomyopathic process may provide a unifying mechanism that associates moderate degrees of PAH and high risk of SD from cardiac causes.

We propose to describe the extent of cardiac involvement in SCA. Specifically, we will (1) describe the LV volume-pressure relations in SCA patients with and without pulmonary hypertension in order to determine how elevated pulmonary pressures are related to dynamic filling properties of the LV; and (2) determine whether cardiac arrhythmias are common in SCA patients with PAH and if they contribute to SD.

Improved understanding of the etiology and mechanisms of SD in SCA may allow the development and testing of therapies for the primary prevention of SD.

ELIGIBILITY:
* INCLUSION CRITERIA FOR RIGHT HEART CATHETERIZATION AND STRESS ECHO:

  1. Either gender, aged greater than 18 years
  2. Diagnosis of sickle cell disease (electrophoretic documentation of SS, SC, or S Beta-thalassemia genotype is required)
  3. Hematocrit greater than 18 % (with an absolute reticulocyte count greater than 100,000/ml)

EXCLUSION CRITERIA FOR RIGHT HEART CATHETERIZATION AND STRESS ECHO:

1. Pregnancy or lactation
2. Known or suspected coronary artery disease
3. Hematocrit less than 18 %: will not be eligible for the study; may return for evaluation at a later date
4. Significant renal insufficiency (patient on hemodialysis or estimated creatinine clearance less than 30% of normal
5. Cerebrovascular accident within the last six weeks
6. New diagnosis of pulmonary embolism within the last three months
7. History of retinal detachment
8. Patients with PAH known to be secondary to other causes, such as systemic lupus erythematosus, other collagen vascular diseases, valvular heart disease, congenital heart disease
9. Poor echo windows
10. Any other condition that would prevent participation in the study (for example HIV infection)

INCLUSION CRITERIA FOR NON-INVASIVE PROCEDURES:

1. Either gender, aged greater than 18 years
2. Diagnosis of sickle cell disease (electrophoretic documentation of SS, SC, or S Beta-thalassemia genotype is required)

EXCLUSION CRITERIA FOR NON-INVASIVE PROCEDURES:

1. Pregnancy or lactation
2. Known or suspected coronary artery disease
3. Significant renal insufficiency (patient on hemodialysis or estimated creatinine clearance less than 30%of normal
4. Cerebrovascular accident within the last six weeks
5. New diagnosis of pulmonary embolism within the last three months
6. History of retinal detachment
7. Patients with PAH known to be secondary to other causes, such as systemic lupus erythematosus, other collagen vascular diseases, valvular heart disease, congenital heart disease
8. Patients who are intolerant of MRI will not undergo cardiac MRI
9. Any other condition that would prevent participation in the study (for example HIV infection)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120
Dates: Start 2005-06-02; Study Completion 2007-10-02

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Suburban Hospital, Bethesda, Maryland
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland

REFERENCES:
- [Background] Charache S. Sickle cells and sudden death. J Lab Clin Med. 1994 Oct;124(4):473-4. No abstract available. PMID 7930871